CLINICAL TRIAL: NCT00194792
Title: Neoadjuvant Complete Hormonal Blockade Followed by Neoadjuvant Chemotherapy for Resectable Hormone Receptor Positive, HER-2/Neu Negative Breast Cancer, A Phase II Study
Brief Title: Hormone Therapy and Combination Chemotherapy Before and After Surgery in Treating Patients With Stage I-IIIA Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Hannah Linden, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6277; NCI-2010-00549 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2005-09-14; First posted 2005-09-19 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Estrogen Receptor-positive Breast Cancer; HER2-negative Breast Cancer; Progesterone Receptor-positive Breast Cancer; Stage I Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; Triptorelin Pamoate; Capecitabine; Methotrexate; merphos; Vinorelbine; Paclitaxel; Taxes; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (hormone therapy and chemotherapy) (Experimental): See detailed description
  Interventions: Drug: exemestane; Drug: triptorelin pamoate; Drug: capecitabine; Drug: methotrexate; Drug: vinorelbine tartrate; Drug: paclitaxel; Procedure: therapeutic conventional surgery; Radiation: radiation therapy; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: exemestane — Given PO
  Other Names: Aromasin; FCE-24304; PNU 155971
Drug: triptorelin pamoate — Given IM
  Other Names: Pamorelin; Trelstar Depot
Drug: capecitabine — Given PO
  Other Names: CAPE; Ro 09-1978/000; Xeloda
Drug: methotrexate — Given IV
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
Drug: vinorelbine tartrate — Given IV
  Other Names: Eunades; navelbine ditartrate; NVB; VNB
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Procedure: therapeutic conventional surgery — Undergo lumpectomy or mastectomy
Radiation: radiation therapy — Undergo radiation therapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well giving hormone therapy together with combination chemotherapy before and after surgery works in treating patients with stage I-IIIA breast cancer. Estrogen can cause the growth of breast cancer cells. Hormone therapy using exemestane and triptorelin pamoate may fight breast cancer by lowering the amount of estrogen the body makes. Drugs used in chemotherapy, such as capecitabine, methotrexate, vinorelbine ditartrate, and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving hormone therapy together with combination chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving these treatments after surgery may kill any tumor cells that remain after surgery

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the pathologic response rate in patients with operable breast cancer treated with a two part, neoadjuvant regimen consisting of complete hormonal blockade (CHB) for 2 weeks followed by four three-week cycles of Xeloda, Methotrexate and Navelbine with continuation of complete hormonal blockade.

SECONDARY OBJECTIVES:

I. To assess the clinical response rate in patients with surgically resectable breast cancer treated with complete hormonal blockade and four three-week cycles of Xeloda, Methotrexate and Navelbine.

II. To assess the toxicity associated with these regimens. III. To assess the relapse rate, overall and disease-free survival in patients with operable breast cancer when treated with neoadjuvant CHB and XMN + CHB followed by adjuvant treatment using XMN or Taxol.

IV. To assess whether the phenotype of breast cancer changes with treatment. V. To assess whether phenotypic changes in breast tumors predict outcome.

OUTLINE:

NEOADJUVANT CHB: Patients receive exemestane orally (PO) daily for 14 weeks. Premenopausal patients also receive triptorelin pamoate intramuscularly (IM) once monthly for 4 months beginning 2 weeks before the initiation of exemestane.

NEOADJUVANT CHEMOTHERAPY: Patients receive capecitabine PO twice daily (BID) on days 1-14 and methotrexate intravenously (IV) and vinorelbine ditartrate IV over 6-10 minutes on days 1, 8, and 15. Treatment repeats every 21 days for 4 courses.

SURGERY: Patients then undergo definitive surgical resection with or without radiation therapy.

ADJUVANT CHEMOTHERAPY: Patients with microscopic complete response (pCR) or disease that has been down-staged to =< 1 cm with no positive nodes receive capecitabine PO BID on days 1-14 and methotrexate IV and vinorelbine ditartrate IV over 6-10 minutes on days 1, 8, and 15. Treatment repeats every 21 days for 4 courses. Patients with down-staged T and 0 or 1 positive node receive paclitaxel IV over 1 hour once weekly for 12 weeks.

ADJUVANT HORMONAL THERAPY: Patients receive hormonal therapy for 5 years.

Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 3 years, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically confirmed, operable ER or PR +, HER2/neu negative, radiographically measurable breast cancer > 1cm (Operable lesions are T1c - T3 and N0 - N2a; histologic confirmation should be by core needle biopsy only)
* Be chemotherapy naive
* Have an ECOG performance status of =< 2
* Be assessed for menopausal status (For study purposes, postmenopausal is defined as: a prior documented bilateral oophorectomy, or a history of at least 12 months without spontaneous menstrual bleeding, or age 60 or older with a prior hysterectomy without oophorectomy, or Age less than 60 with a prior hysterectomy without oophorectomy [or in whom the status of the ovaries is unknown], with a documented FSH level demonstrating confirmatory elevation in the postmenopausal range for the lab)
* All premenopausal patients must have a baseline FSH and LH
* ANC >= 1,500
* Platelet count >= 100,000
* Serum creatinine =< 1.5 x IULN
* Estimated creatinine clearance > 50 ml/min
* Have staging studies and tumor assessment prior to registration
* Bone density exam must be done within the first 3 months of complete hormonal blockade
* Have a negative pregnancy test within seven days prior to registration if of childbearing potential
* Be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study specific screening procedures

Exclusion Criteria:

* Primary tumor =< 1 cm, not measurable; inflammatory disease
* Pregnant or lactating; women of childbearing potential with either a positive or no pregnancy test at baseline are excluded (Women of childbearing potential who are not using a reliable and appropriate contraceptive method are excluded; patients must agree to continue contraception for 30 days from the last study drug administration)
* Prior unanticipated severe reaction to fluoropyrimidine therapy, or known sensitivity to 5-fluorouracil
* Previous enrollment in an investigational drug study within the last 4 weeks
* Evidence of distant metastatic disease
* Prior chemotherapy or hormonal therapy for breast cancer
* Prior malignancy other than adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, other stage I or II cancer from which the patient has been disease free for at least 5 years
* History of uncontrolled seizures, central nervous system disorders, or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance with oral drug intake
* Any other life-threatening illness (e.g. serious, uncontrolled concurrent infection or clinically significant cardiac disease - congestive heart failure, symptomatic coronary artery disease, cardiac arrhythmia not well controlled with medication or myocardial infarction
* Major surgery within four weeks of the start of study treatment without complete recovery
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome
* Known, existing uncontrolled coagulopathy
* Unwillingness to give informed consent
* Unwillingness to participate or inability to comply with the protocol for the duration of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2005-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Linden, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Hormone Therapy and Chemotherapy)
Started | 28
Completed | 27
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Hormone Therapy and Chemotherapy)
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 55 [35 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 26
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Response
Description: Defined as a > 50% decrease in sum of the products of the perpendicular diameters of bidimensionally measurable disease.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Hormone Therapy and Chemotherapy)
Number analyzed (Participants) | 27
Participants | 19

2. Primary Outcome: Number of Participants With Microscopic Pathologic Complete Response and Macroscopic Pathologic Complete Response
Description: Defined as no evidence of microscopic invasive tumor at the primary site or in the regional lymph nodes at the time of definitive surgical resection and the examining pathologist cannot identify gross residual tumor mass in the surgical specimen.
Time Frame: From date of treatment start to surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Hormone Therapy and Chemotherapy)
Number analyzed (Participants) | 27
Participants | 0

3. Primary Outcome: Disease-free Survival
Description: Kaplan-Meier estimate assessed at 5 years
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: disease free survival probability
Arm/Group | Treatment (Hormone Therapy and Chemotherapy)
Number analyzed (Participants) | 27
disease free survival probability | 0.76 [0.61 to 0.95]

4. Primary Outcome: Overall Survival
Description: From the start of protocol therapy until the date of death from any cause or the last date the patient was known to be alive. Kaplan-Meier estimate assessed at 5 years.
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | Treatment (Hormone Therapy and Chemotherapy)
Number analyzed (Participants) | 27
survival probability | 0.88 [0.76 to 1]

5. Primary Outcome: Quantification of All Grade 2, 3, 4 Adverse Events or Fatal Toxicities
Description: Count of all incidences of grade 2, 3, 4 adverse events and fatal toxicities
Time Frame: Monthly during neoadjuvant treatment and then 6 months following treatment (including surgery)
Measure: Number; unit: events
Arm/Group | Treatment (Hormone Therapy and Chemotherapy)
Number analyzed (Participants) | 27
events
  Grade 2 | 80
  Grade 3 | 12
  Grade 4 | 0
  Fatal toxicity | 0

6. Primary Outcome: Number of Participants With Dose Reduction, Treatment Interruption, or Treatment Discontinuation
Description: Count of patients with dose reduction, treatment interruption, or treatment discontinuation.
Time Frame: During adjuvant and neoadjuvant chemotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Hormone Therapy and Chemotherapy)
Number analyzed (Participants) | 27
Participants
  Adjuvant therapy | 1
  Neoadjuvant therapy | 11

7. Secondary Outcome: Correlation of Molecular Markers With Response, Time to Progression, and Survival
Time Frame: Weekly during CHB and XMN and pacitaxel
Population: Molecular marker data was not collected for this cohort and thus not possible to report results for this outcome.
Arm/Group | Treatment (Hormone Therapy and Chemotherapy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment (Hormone Therapy and Chemotherapy)
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 23/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Hormone Therapy and Chemotherapy) (N=27)
High Blood Pressure (Vascular disorders) | 2
Fatigue (General disorders) | 17
Nausea (Gastrointestinal disorders) | 16
Dysgeusia (Gastrointestinal disorders) | 4
Fever (General disorders) | 4
SGOT Increased (Investigations) | 9
SGPT Increased (Investigations) | 10
Albumin Decreased (Investigations) | 5
Potassium Decreased (Investigations) | 7
Anxiety (Psychiatric disorders) | 4
Diarrhea (Gastrointestinal disorders) | 7
Alopecia (Skin and subcutaneous tissue disorders) | 3
Mucositis (GI) (Gastrointestinal disorders) | 2
Mucositis (Oral) (Gastrointestinal disorders) | 6
Neutrophil Count Decreased (Investigations) | 14
Alkaline Phosphatase Increased (Investigations) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Insomnia (Psychiatric disorders) | 6
Heartburn (Gastrointestinal disorders) | 2
Hemoglobin Decreased (Investigations) | 16
White Blood Cells Decreased (Investigations) | 18
Depression (Psychiatric disorders) | 7
Pain (arm) (General disorders) | 2
Hot Flashes/Night Sweats (Vascular disorders) | 14
Pain (neck & jaw) (General disorders) | 2
Pain (back) (General disorders) | 4
Constipation (Gastrointestinal disorders) | 5
Headache (Nervous system disorders) | 4
Pain (subcostal) (General disorders) | 3
Pain (abdominal) (Gastrointestinal disorders) | 3
Dry Skin (hands) (Skin and subcutaneous tissue disorders) | 2
Hematocrit Decreased (Investigations) | 2
Hypocalcemia (Investigations) | 3
Joint Pain/Muscle Aches (General disorders) | 5
Amenorrhea (Reproductive system and breast disorders) | 2
GI Upset/Reflux (Gastrointestinal disorders) | 2
Sodium Decreased (Investigations) | 3
Hand Foot Syndrome (Skin and subcutaneous tissue disorders) | 4
Common Cold (Respiratory, thoracic and mediastinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 2
Rash (Eczema) (Skin and subcutaneous tissue disorders) | 2
Lactate Dehydrogenase Increased (Investigations) | 7
Glucose Increased (Investigations) | 3
Pain (bone) (Musculoskeletal and connective tissue disorders) | 3
Yeast Infection (vaginal) (Reproductive system and breast disorders) | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 4
SOB with activity (Respiratory, thoracic and mediastinal disorders) | 3
UTI (Renal and urinary disorders) | 3
Hyperpigmentation (lymphs) (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes